CLINICAL TRIAL: NCT01880398
Title: Case Study of Fistula in Ano Managed by Kshar Sutra, Para Surgical Procedure
Brief Title: Management of Fistula in Ano by Kshar Sutra, Para Surgical Procedure.
Acronym: Bhagandar
Status: Completed | Type: Observational
Sponsor: Government Ayurved College and Hospital (Other Government)
Responsible Party: Principal Investigator, Dr.Nita Mahadevrao Kedar, Associate professor, Government Ayurved College and Hospital
Other Study IDs: 2468
Record Dates: First submitted 2013-06-09; First posted 2013-06-19 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Fistula in Ano
Keywords: FIstula in ano; Bhagandar
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Kshar Sutra: The Kshar Sutra was a standard medicated thread smeared with Kshar of Apamarga (Achyranthus aspera), Shnuhi (Eforbia Nerrifolia) which has quality of cutting and Haridra(Curcuma Longa) which is used as a antiseptic. The ph value of the thread thus prepared was determined and its sterilization effected by ultraviolet radiation. The alkalinity of Kshar Sutra was 9.2ph.
  Interventions: Other: Kshar Sutra

INTERVENTIONS:
Other: Kshar Sutra — The Kshar Sutra was a standard medicated thread smeared with Kshar of Apamarga (Achyranthus aspera), Shnuhi (Eforbia Nerrifolia) which has quality of cutting and Haridra(Curcuma Longa) which is used as a antiseptic. The ph value of the thread thus prepared was determined and its sterilization effected by ultraviolet radiation. The alkalinity of Kshar Sutra was 9.2ph.
  Other Names: Medicated Thread

SUMMARY:
Background: Fistula in ano is one of the most common diseases of the ano rectal region. Treatment of Fistula in ano has puzzled the medical fraternity due to its complex nature. Commonly prevalent surgical treatment for anal Fistula, that is "Fistulectomy" does not provide successful cure for the disease, post operative complications and recurrences being common. Acharya Sushruta an ancient Indian Surgeon has described in his text ' Sushruta Samhita' about an ancient Ayurvedic technique of medicated thread called Ksharsutra treatment for Bhagandara ( Fistula in ano). Treatment of anal Fistula (Bhagandara)and Nadi-Vrana(Sinus) with Ksharsutra was practiced by Sushruta (1000-600B.C.) .

Hypothesis: Aycharya Sushruta advocated Kshar Sutra therapy in Fistula in ano and in various types of Fistula.

DETAILED DESCRIPTION:
A 48 years old female patient, came with complaints of painful discharging boil at left side of Perianal region with pain.

She gave a surgical history of incision and drainage for gluteal abscess done in before four month. On local examination Patient had discharging sinus at 3 o' clock position on left side of Perianal region. Before planning the treatment other aetiologies were ruled out.

Diagnosis was confirmed by Fistulogram, suggestive of high anal fistula with internal opening in the anal canal. Under spinal anaesthesia probing was done. Internal opening of Fistula was confirmed by injecting Methylene Blue dye through external opening. The track was directed upward in the anal canal without any tributaries. Length of the tract was 9cm.

Then Kshar Sutra was tied covering the entire underlying track for cutting and healing under all aseptic precaution. The patient was discharged on the next day of procedure. The Kshar Sutra was changed weekly. To promote healing and to reduce pain and inflammation oral antibiotics, anti-inflammatory medicine were also prescribed.

The total period of Kshar Sutra treatment was 5 month. The Kshar Sutra was a standard medicated thread smeared with Kshar of Apamarga (Achyranthus aspera), Shnuhi (Eforbia Nerrifolia) which has quality of cutting and Haridra(Curcuma Longa) which is used as a antiseptic. The ph value of the thread thus prepared was determined and its sterilization effected by ultraviolet rediation. The alkalinity of Kshar Sutra was 9.2ph.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Fistula in ano without tributeries.

Exclusion Criteria:

* Multiple fistula and associated ano rectal conditions

Min Age: 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Government Ayurved Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of Kshar sutra in Fistula in ano | 5month
  Cutting and healing of the Fistula track.

SECONDARY OUTCOMES:
Recurrence of Fistula in ano | 1year
  By observing patient for 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Nita M Kedar, M.S.(Ayu), Principal Investigator — Government Ayurved Hospital
Locations (1):
- Government Ayurved Hospital, Nagpur, Maharashtra, India